CLINICAL TRIAL: NCT05668299
Title: Determining the Appropriate Setting of an Automated Secretion Removal Technology (TrachFlush) Danish Title: Bestemmelse af Den Optimale Indstilling for en Teknologi Til Automatisk Fjernelse af Luftvejssekret (Trachflush)
Brief Title: Determining the Appropriate Setting of an Automated Secretion Removal Technology (TrachFlush)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitalsenheden Vest (Other)
Collaborators: Viborg Regional Hospital (Other); Herning Hospital (Other); Aalborg University (Other)
Responsible Party: Principal Investigator, Anne Højager Nielsen, Head of Research, Hospitalsenheden Vest
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEK protocol 76288
Record Dates: First submitted 2022-12-12; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Mechanical Ventilation Complication; Intubation Complication
Keywords: Mechanical Ventilation; Suctioning; Critically ill patients; Secretion

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TrachFlush group (Experimental): Patients in this arm received the intervention.
  Interventions: Device: TrachFlush

INTERVENTIONS:
Device: TrachFlush — See detailed description previously entered.

SUMMARY:
Using a new device, the TrachFlush, the aim of this pilot study is to investigate whether secretions can be removed at the patient's current ventilator settings, or whether pressures and durations considered at the maximal end of clinical practice are required, so as to push secretions around the cuff. The study is a pilot study to investigate the settings required to ensure clinical efficacy of the technology, prior to large scale clinical studies.

DETAILED DESCRIPTION:
Design:

Prospective, non-controlled, pilot study of the TrachFlush© technology on 20 patients, mechanically ventilated in the intensive care unit.

Study procedure This study is designed to evaluate whether the TrachFlush technology the symptoms associated with need of tracheal suctioning, when applied at the patient's current ventilator settings, or following a change in ventilator settings to the maximal inspiratory pressure and time acceptable in clinical practice. Figure 2 illustrates the protocol procedure. Patients will be studied during mechanical ventilation when on pressure control or pressure support mode. When recruited, and on clinical need for suctioning, the patient will be evaluated to see if they are eligible for the TrachFlush procedure. If the patient is on a volume regulated mode; has an inspiratory time < 1 second; has a value of positive end expiratory pressure >15 cmH2O; has a PaO2 (arterial partial pressure of oxygen)/FiO2 (fraction of inspired oxygen) ratio lower that 100 mmHg, i.e. indicative of severe ARDS (acute respiratory distress syndrome); or has tachycardia defined as >120 bpm then the patient will be considered ineligible for the procedure. As such, the patient will be considered again on the next clinical need for suctioning. On detection of a clinical need for suctioning, and when the patient is eligible for the TrachFlush procedure, the reason for suctioning will be documented - as inadequate oxygenation, rising ventilation pressures with disturbing ventilation pressure waveforms, or audible sounds of secretions. The TrachFlush procedure will then be performed following the 5 steps described below:

1. Ventilator settings for inspiratory pressure, positive end expiratory pressure and, for control mode, respiratory rate will be maintained at current clinical values.
2. The TrachFlush "button" will be pressed three times over a period of 1 minute, allowing 3 cuff deflations and inflations during 3 non-consecutive inspirations. As the procedure is rapid, no pre-oxygenation will be performed. SpO2 (oxygen saturation) will be monitored continuously and oxygen flushing applied immediately, should oxygenation deteriorate.
3. Following this procedure, clinical indications towards the need of suctioning will be re-evaluated and recorded, with two possible outcomes as evaluated by the investigator at the bedside.

   i. Success - Clinical state is such that endotracheal suctioning is no longer required.

   ii. Failure - Clinical state has not improved sufficiently. For case 1 suctioning is not performed, suctioning of the mouth is permitted. For case 2, ventilator settings are adjusted to a maximal safe level for the short duration, i.e.

   PEEP(positive end expiratory pressure) and pressure support or pressure control will be increased such that the sum of these, i.e. the peak pressure is 30 cmH20. In doing so, PEEP will not be > 15 cmH2O.

   For control mode ventilation, if respiratory rate is higher than 10 breaths per minute, this will be reduced to 10, to allow increase in inspiratory time. In addition, the TrachFlush device will be set to deliver the cuff deflation and inflation over a longer period, allowing increased time to remove secretions. This setting can be performed directly on the device and will be set to be 100 ms lower than the inspiratory time achieved with a respiratory rate of 10, allowing for full cuff deflation and inflation within this period.

   For either of these situations, if current settings are already at maximal pressure and minimal respiratory frequency, the protocol will move to step 5, with that step recorded as a failure.
4. Following modification of ventilator settings, the TrachFlush "button" will be pressed three times over a period of 1 minute, allowing 3 cuff deflations and inflations during 3, non-consecutive inspirations, as previously described.
5. Following this procedure, clinical indications of the need for suctioning will be re-evaluated and recorded, with two possible outcomes.

   i. Success - Clinical state is such that endotracheal suctioning is no longer required. Suctioning of the mouth is permitted. ii. Failure - Clinical state has not improved sufficiently.
6. Ventilator settings will be returned to baseline values and following failure of the TrachFlush procedure, clinical suctioning will be performed if necessary and in accordance with normal clinical practice.

All tasks will be performed by the research team associated with the project. To assess intra-patient variability, the above procedure will be performed 3 times on the same patient, for three different occasions where there is a need for airway suctioning. As an average of 3 suctions are performed routinely per patient per day, it is expected that this study will take 1 day with a maximum of 2 days per patient.

ELIGIBILITY:
Inclusion Criteria:

* Orally intubated and mechanically ventilated
* Patients for whom it is expected that secretions will be present during their ventilation period, as assessed by clinical evaluation.

Exclusion Criteria:

* Admission due to tracheal damage, e.g. inhalation trauma.
* Severe ARDS (acute respiratory distress syndrome), indicated by a PaO2/FiO2 ratio lower than 100 mmHg or PEEP > 15 cmH2O.
* Circulatory instability indicated by use of vasopressor (Norepinephrine) >0.1 micro gm/kg/min, heart rate >120, arrhythmia other than atrial fibrillation.
* Patients with agitated delirium.
* Mechanical ventilation via tracheostomy
* Mechanical ventilation is provided with a mask or other non-invasive means
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Ability to remove secretion from tube | Immediately after the procedure.
  Success - clinical state is such that endotracheal suctioning is no longer required; Failure - clinical state has not improved sufficiently.

SECONDARY OUTCOMES:
Procedures performed using increased settings. | Immediately after the procedure
  Number of patients needing increased ventilator settings.
Patient comfort | Immediately after the procedure
  Evaluated using the Critical-care Pain Observation Tool (CPOT), a scale from 0-8 points, higher values indicating higher levels of pain/distress in the mechanically ventilated patient.
Hypoxia | Immediately after the procedure
  Indicated as more than 10% decrease of SpO2.

CONTACTS AND LOCATIONS:
Overall Officials: Nilanjan Dey, MD, Principal Investigator — Gødstrup Hospital
Locations (2):
- Denmark (2):
  - Regional Hospital Herning, Herning, Central Jutland
  - Regional Hospital Viborg, Viborg, Central Jutland

IPD SHARING:
Plan to Share IPD: No
The investigators do not have permission to share individual participant data.

REFERENCES:
- [Background] Turner JS, Briggs SJ, Springhorn HE, Potgieter PD. Patients' recollection of intensive care unit experience. Crit Care Med. 1990 Sep;18(9):966-8. doi: 10.1097/00003246-199009000-00012. PMID 2394120
- [Background] Granja C, Lopes A, Moreira S, Dias C, Costa-Pereira A, Carneiro A; JMIP Study Group. Patients' recollections of experiences in the intensive care unit may affect their quality of life. Crit Care. 2005 Apr;9(2):R96-109. doi: 10.1186/cc3026. Epub 2005 Jan 31. PMID 15774056
- [Background] Maggiore SM, Lellouche F, Pignataro C, Girou E, Maitre B, Richard JC, Lemaire F, Brun-Buisson C, Brochard L. Decreasing the adverse effects of endotracheal suctioning during mechanical ventilation by changing practice. Respir Care. 2013 Oct;58(10):1588-97. doi: 10.4187/respcare.02265. Epub 2013 Mar 6. PMID 23466423
- [Background] Efrati S, Deutsch I, Antonelli M, Hockey PM, Rozenblum R, Gurman GM. Ventilator-associated pneumonia: current status and future recommendations. J Clin Monit Comput. 2010 Apr;24(2):161-8. doi: 10.1007/s10877-010-9228-2. Epub 2010 Mar 17. PMID 20237830
- [Background] Li J, Zong Y, Zhou Q, Dai H, Wang C. Evaluation of the Safety and Effectiveness of the Rapid Flow Expulsion Maneuver to Clear Subglottic Secretions in Vitro and in Vivo. Respir Care. 2017 Aug;62(8):1007-1013. doi: 10.4187/respcare.05348. Epub 2017 Apr 4. PMID 28377403
- [Background] Zanella A, Florio G, Rezoagli E, Pastore M, Cadringer P, Biancolilli O, Carlesso E, Scaravilli V, Ristagno G, Pesenti AM. An Artificial Cough Maneuver to Remove Secretions From Below the Endotracheal Tube Cuff. Respir Care. 2019 Apr;64(4):372-383. doi: 10.4187/respcare.06076. Epub 2019 Jan 8. PMID 30622174
- [Background] Gelinas C, Fillion L, Puntillo KA, Viens C, Fortier M. Validation of the critical-care pain observation tool in adult patients. Am J Crit Care. 2006 Jul;15(4):420-7. PMID 16823021
- [Background] Frandsen JB, O'Reilly Poulsen KS, Laerkner E, Stroem T. Validation of the Danish version of the Critical Care Pain Observation Tool. Acta Anaesthesiol Scand. 2016 Oct;60(9):1314-22. doi: 10.1111/aas.12770. Epub 2016 Jul 29. PMID 27468726